CLINICAL TRIAL: NCT03584841
Title: Implementation of a Non-invasive Version of the Imaging β-adrenergic-dependent Sweat Secretion Test: Value for Diagnosis and Efficacy of Target Therapies for Cystic Fibrosis
Brief Title: Implementation of a Non-invasive Version of the Imaging β-adrenergic-dependent Sweat Secretion Test
Acronym: BUBBLE TEST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015/04MAI/231
Record Dates: First submitted 2018-05-27; First posted 2018-07-12 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Mucoviscidosis Involving the Lung
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: Intervention Model: Three Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with mucoviscidosis (Experimental): For patients with cystic fibrosis: clinically stable, all genotypes included.
  Interventions: Diagnostic Test: Iontophoresis sessions in forearm of subjects with pilocarpine
- Parents of patients with confirmed diagnosis of mucoviscidosis (Experimental): The parents are heterozygous subjects
  Interventions: Diagnostic Test: Iontophoresis sessions in forearm of subjects with pilocarpine
- Healthy volunteers (Active Comparator)
  Interventions: Diagnostic Test: Iontophoresis sessions in forearm of subjects with pilocarpine

INTERVENTIONS:
Diagnostic Test: Iontophoresis sessions in forearm of subjects with pilocarpine — The test with two iontophoresis sessions is performed in a forearm of subjects. Pilocarpine is applied during the first iontophoresis session to evoke cholinergic-induced sweat secretion. Atropine, isoprenaline and aminophylline are applied during the second iontophoresis session, to block the cholinergic component and to evoke β-adrenergic-induced sweat secretion.

SUMMARY:
The goal of this study is to implement a non-invasive version of the sweat secretion test based in visualization of sweat glands following β-adrenergic stimulation of sweat. Specifically, the trial will evaluate the relative response of sweat glands to β-adrenergic and cholinergic stimulation among participants with CF, heterozygous and matched control subjects

ELIGIBILITY:
Inclusion Criteria:

* For patients with cystic fibrosis: clinically stable, all genotypes included.
* For healthy volunteer and heterozygous subjects: 18 years and older.

Exclusion Criteria:

* Corticosteroids, anti-leukotriene therapy, unstable clinical status, <40% FEV1.
* Current pregnancy or breastfeeding.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-03-31 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Ratio between the β-adrenergic/cholinergic rate | up to 30 minutes
  The ratio between the β-adrenergic/cholinergic rate (nL/min) of droplets of sweat is calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
There is no plan now